CLINICAL TRIAL: NCT04493749
Title: Clinical Performance of Withings Move ECG Software for Atrial Fibrillation Detection
Acronym: ECG-SW1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A013-58-49
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- atrial fibrillation (AF): Patients diagnosed with AF during reference ECG
  Interventions: Diagnostic Test: ECG measurement
- sinus rhythm (SR): Patients diagnosed with SR during reference ECG
  Interventions: Diagnostic Test: ECG measurement

INTERVENTIONS:
Diagnostic Test: ECG measurement — Simultaneous recording of a single-lead ECG signal with the Withings Move ECG and ECG signal for the reference 12-lead ECG

SUMMARY:
Withings Move ECG watch is designed to record ECG and detect automatically atrial fibrillation. The aim of this study is to validate the performance of Move ECG watch to detect atrial fibrillation compared to a reference 12-lead ECG.

DETAILED DESCRIPTION:
Patients with atrial fibrillation are included in hospitals. On each patient, ECG with Move ECG and the reference 12-lead ECG are recorded simultaneously. Both records are then reviewed by independent cardiologists to assess

1. The presence or absence of atrial fibrillation
2. if waveforms of ECG recorded with Move ECG compared with the reference.

ELIGIBILITY:
Inclusion Criteria:

* male or female who are 18 years or older
* Subject who signed the written informed consent form

Exclusion Criteria:

* Vulnerable subject with regard to regulations
* Pregnant, parturient or breastfeeding woman,
* Subject who is deprived of liberty by judicial, medical or administrative decision,
* Underage subject,
* Legally protected subject, or subject who is unable to sign the written informed consent form,
* Subject who is not beneficiary or not affiliated to a social security scheme,
* Subject within several of the above categories,
* Subject who refused to participate in the study,
* Subject in physical incapacity to wear a wrist-worn watch
* Subject with electrical stimulation by pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in and out patients from cardiology services
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the automatic classification in AF by Move ECG single-lead ECG against reference 12-lead ECG | 1 year
  sensitivity from the 2x2 confusion matrix AF vs 'non-AF'

SECONDARY OUTCOMES:
Comparability of ECG waveforms from single strip of Move ECG vs Lead-1 of reference 12-lead ECG | 1 year
  Visibility and polarity of P waves, QRS complex and T waves + length of QT interval, QRS width and PR interval + heart rate
Safety of use of Move ECG | 1 year
  Frequency of adverse event appearance

CONTACTS AND LOCATIONS:
Overall Officials: Julien Nahum, Principal Investigator — Centre Cardiologique du Nord
Locations (3):
- France (3):
  - Institut Cœur Paris Centre Turin, Paris, Île-de-France Region
  - Hopital Europeen Georges Pompidou, Paris, Île-de-France Region
  - Centre Cardiologique du Nord, Saint-Denis, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No